CLINICAL TRIAL: NCT07098507
Title: Real-world Integration of De-Escalation in Axillary Surgery for Postmenopausal, Early Stage HR+HER2- Breast Cancer Patients
Brief Title: De-escalation in Axillary Surgery for Early-stage Breast Cancer
Acronym: RIDES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Ana Car Peterko, General Surgeon and surgical oncologist, FEBS (breast surgery), CEBS, Clinical Hospital Center Rijeka
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2170-29-02/15-25-2
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Omitting Sentinel Lymph Node Biopsy in Early-stage Breast Cancer
Keywords: breast cancer; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (NO-SLNB) (Experimental): Sentinel lymph node biopsy will be omitted for all participants
  Interventions: Procedure: omission of sentinel lymph node biopsy
- Standard of care (SLNB) (Active Comparator): Standard of care treatment (SLNB) will be performed in all participants
  Interventions: Procedure: sentinel lymph node biopsy

INTERVENTIONS:
Procedure: sentinel lymph node biopsy — As sentinel lymph node biopsy is still a standard of care in early-stage breast cancer surgery, it represents the intervention in the standard of care arm
  Arms: Standard of care (SLNB)
Procedure: omission of sentinel lymph node biopsy — omission of sentinel lymph node biopsy is the intervention in the experimental arm
  Arms: Experimental arm (NO-SLNB)

SUMMARY:
The goal of this clinical trial is to determine if the omission of sentinel lymph node biopsy is safe for early-stage breast cancer patients in our institution (Clinical Hospital Centre Rijeka).

Targeted group are postmenopausal patients, older than 55 years, diagnosed with hormone-receptor-positive breast cancer, with primary tumour less than 3 cm and unaffected axilla on clinical exam and axillary ultrasound.

The main questions we aim to answer are:

* if this treatment de-escalation affects patient oncological outcomes (cancer recurrence)?
* if this treatment de-escalation affects patient clinical outcomes (early and late complications related to axillary surgery)?
* if this omission of pathological examination of sentinel lymph node affects recommendations on postoperative treatments (irradiation and systemic therapy)? Researchers will compare outcomes between participants submitted to sentinel lymph node biopsy and participants in whom the procedure is omitted to answer those questions.

Participants will be asked to:

* decide in which group they wish to participate
* visit the clinic for checkups and tests once every 6 months in first two years and yearly thereafter up to 5 years

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed hormone receptor positive, HER2 negative invasive breast cancer or DCIS with microinvasion, histologically confirmed, in postmenopausal patients older than 55 years, with primary tumour up to 3 cm and uninvolved axillary lymph nodes on clinical examination and on axillary ultrasound performed in Clinical Hospital Centre Rijeka. Patients should be eligible for breast conserving surgery and adjuvant whole breast irradiation.

Exclusion Criteria:

* Patients younger than 55 years of age and/or premenopausal, with cN1-3 status (confirmed cytologically or histologically), or with multiple suspicious lymph nodes on axillary ultrasound, regardless of cytological/histological confirmation.
* Patients diagnosed with pure breast carcinoma in situ (DCIS) without focal invasion
* Patients with tumour larger than 3 cm or with cT4 status, with de novo metastatic disease
* Patients with a breast cancer of HER2+ or triple-negative immunophenotype
* Patients who have received any type of neoadjuvant systemic therapy before surgery and those who have a previous personal history of invasive breast cancer
* Patients with extensive multifocal or multicentric breast cancer, patients scheduled for mastectomy, partial breast irradiation or who refuse recommended adjuvant systemic oncological treatment
* Patients who do not wish to participate in a clinical trial

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2033-09-10 (Estimated); Study Completion 2033-09-10 (Estimated)

PRIMARY OUTCOMES:
Isolated regional recurrence free survival | 5 years
  Isolated axillary lymph node recurrence free interval (time from surgery until axillary lymph node recurrence, provided that axillary recurrence is the first and only recurrence)
Disease free survival | 5 years
  Cancer recurrence-free interval (time from surgery until any recurrence)

SECONDARY OUTCOMES:
Isolated regional recurrence rate | 5 years
  Rate of isolated recurrence in axillary lymph nodes
Any invasive recurrence rate | 5 years
  Overall recurrence rate (in breast, axillary lymph nodes or distant sites)
Rate of adjuvant chemotherapy recommendation in standard and experimental arm | 5 years
  Differences in adjuvant chemotherapy recommendation between standard and experimental arm.
Rate of adjuvant regional nodal irradiation in standard and experimental arm | 4 years
  Difference in regional nodal irradiation rate between standard and experimental arm
Rate of early postoperative complications in axilla in standard arm | 3 years (accrual period)
  Rate of haematoma, seroma and wound infection in axilla after SLNB
Rate of late complications of axillary surgery in standard arm | 5 years
  Rate of arm paraesthesia, decreased range of motions in shoulder and arm lymphedema

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Centre Rijeka, Rijeka, Croatia